CLINICAL TRIAL: NCT01660516
Title: Effect of Black Tea Consumption on Endothelial Function and Ischaemia-reperfusion Injury in Humans
Brief Title: Effect of Tea on Endothelial Function and Ischaemia-reperfusion Injury
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: TEA-IRI; Tea-IR-Injury-FMD (Other: Radboud University Nijmegen Medical Centre)
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2012-07

CONDITIONS: Ischaemia Reperfusion Injury
Keywords: Camellia sinensis; flavonoids; cardiovascular risk; flow mediated dilation
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tea: Black tea ingestion

SUMMARY:
Tea consumption may impact upon the decrease in endothelial function after IR-injury. However, no previous study directly examined the potential of tea to impact upon the change in endothelial function after IR-injury.

The investigators hypothesize that tea consumption counteracts endothelial damage in response to ischaemia reperfusion injury in healthy humans.

DETAILED DESCRIPTION:
Rationale: Occlusion of an artery (causing ischemia) is a frequently reported condition, e.g. myocardial infarction, cerebral infarction or during organ transplantations. The period of ischemia will be followed by reperfusion (possibly after an operation). The ischaemic period as well as the reperfusion are both associated with damage to the tissue, including the endothelium. It is hypothesised that production of oxidative stress and reduced NO bioactivity (through increased reactive oxygen production) during ischaemia and reperfusion is involved in the development of tissue damage to the endothelium. Interventions that can prevent or attenuate endothelial dysfunction in response to ischemia-reperfusion (IR)-injury have a potential clinical relevance to prevent (complications of) cardiovascular disease.

Several studies have examined the effect of tea consumption on the endothelial function. These studies demonstrated a dose-dependent improvement of tea to improve endothelial function in healthy and diseased humans, possibly through the vasoactive effects of flavonoids, which may involve increased nitric oxide bioactivity and inhibition of NADPH oxidase. Based on the ability of flavonoids to decrease (the impact of) oxidative stress, tea consumption may also impact upon the decrease in endothelial function after IR-injury. However, no previous study directly examined the potential of tea to impact upon the change in endothelial function after IR-injury.

Objective: To examine whether tea consumption counteracts endothelial damage in response to ischaemia reperfusion injury in healthy humans.

Main study parameters: Change in endothelial function (measured with flow mediated dilation) after ischaemia reperfusion injury (induced by 20 minutes ischemia and 20 min reperfusion) with and without precedence of tea consumption.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Non-invasive cuff occlusion is used to examine endothelial function (5-minute ischaemia) and produce the stimulus that induces ischaemia-reperfusion injury (20-minute ischaemia). This repeated cuff inflation is non-invasive and not associated with a health risk for the subject. Tea consumption is safe and, most likely, daily routine for most participants. The only difference is that this study will monitor and instruct participants regarding their tea consumption in the week preceding the tests. The volunteers will not benefit directly from participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers : age 18-60
* All subjects: written informed consent

Exclusion Criteria:

* Smoking
* History of any cardiovascular disease
* Hypertension (in supine position: systole >140 mmHg, diastole >90 mmHg)
* Diabetes Mellitus
* Hyperlipidaemia (fasting total cholesterol >6.5 mmol/L)
* Chronic use of medication known to interfere with the cardiovascular system
* Professional athletes
* Alcohol consumption >14 units/week
* BMI >30 kg/m2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty-one volunteers, aged between 30 and 70 years, were included in our study. All subjects were healthy and free of (a history of) cardiovascular disease or obesity (BMI >30 kg/m2). Individuals were excluded if they reported a chronic or acute disease, including any kind of metabolic abnormality (such as diabetes mellitus) or cardiovascular disease. Habitual smokers (n=3) were instructed to withdraw from smoking on the day of testing. To further avoid confounding factors, the investigators also excluded individuals reporting daily intense sporting activities (>10 h/w), and/or were treated with a diet due to any reason.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change in Endothelial Function after ischaemia reperfusion injury | three weeks
  Change in endothelial function (measured with flow mediated dilation) after ischaemia reperfusion injury (induced by 20 minutes ischemia and 20 min reperfusion) with and without precedence of tea consumption

SECONDARY OUTCOMES:
Change in baseline flow mediated dilation after water/tea consumption | three weeks
  Change in baseline flow mediated dilation after water/tea consumption

CONTACTS AND LOCATIONS:
Overall Officials: Dick Thijssen, Dr., Principal Investigator — Radboud University Medical Centre Nijmegen; Maria Hopman, Prof. Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands